CLINICAL TRIAL: NCT06142513
Title: The Effect of Obesity Hypoventilation Syndrome on Exercise Capacity, Peripheral Muscle Strength, and Quality of Life in Obese Individuals
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proffesor, Istanbul University
Other Study IDs: 2023-1/GAslan
Record Dates: First submitted 2023-11-11; First posted 2023-11-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Obesity Hypoventilation Syndrome; Obesity; Hypoventilation; Respiration Disorders; Sleep Disorder; Breathing-Related
Keywords: Obesity; Obesity Hypoventilation Syndrome; Exercise Capacity; Quality of Life; Peripheral Muscle Strength
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Obesity; Hypoventilation; Respiration Disorders; Sleep Wake Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Grup I: Subjects with obesity hypoventilation syndrome (30 < body mass index < 45 kg/m2)
  Interventions: Other: Assessment
- Grup II: Age and sex-matched obese subjects (30 < body mass index < 45 kg/m2) with low risk of obstructive sleep apnea (STOP-BANG score < 3)
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Between December 2023 and June 204, 46 volunteer participants aged 18 years and older who met the inclusion criteria and were followed up at Istanbul University, Istanbul Faculty of Medicine, Department of Chest Diseases and Istanbul Faculty of Medicine, Department of Internal Medicine were included in the project. Participants' body composition, comorbidities, exercise capacity, peripheral muscle strength, sleep quality and quality of life were assessed.

SUMMARY:
Obesity Hypoventilation Syndrome(OHS) is a disease characterized by daytime hypercapnia and sleep-disordered breathing without other causes of hypoventilation in individuals with a body mass index above 30 kg/m2. Sources state that obesity is at the basis of the metabolic changes seen in individuals with OHS. Obesity, together with cardiovascular system complications, lung volumes, work of breathing and sleep quality, creating the basis for respiratory problems. In addition, sedentary lifestyle habits, which are common in obese individuals, cause negative effects on exercise capacity and peripheral muscle strength. It has been shown in the literature that decreased exercise capacity due to obesity strongly interacts with the risk of all-cause mortality. As a result of obesity and all this negative picture, impaired emotional state and decreased quality of life are observed in individuals. Numerous studies have shown that obese individuals generally have a low level of physical activity, there is a decrease in peripheral muscle strength, obese individuals are at risk for sleep-related respiratory problems and health-related quality of life is often negatively affected in obese individuals. With these studies, the effects of obesity on individuals have been evaluated with objective evaluation methods. However, the same cannot be said for OHS. It is not clear how exercise capacity, peripheral muscle strength and quality of life parameters, which are known to be negatively affected by obesity, are affected in individuals with OHS. Based on this point, this study aims to investigate whether OHS has an additional effect on exercise capacity, peripheral muscle strength and quality of life in addition to obesity.

DETAILED DESCRIPTION:
Patients with Obesity Hypoventilation Syndrome who are followed up in Istanbul University, Istanbul Faculty of Medicine, Department of Chest Diseases and obese individuals who are followed up in Istanbul University, Istanbul Faculty of Medicine, Department of Internal Diseases and who are in the low risk group according to stop bang evaluation will be included in the study. The data of individuals diagnosed with OHS and obese individuals will be compared. The study will be conducted in accordance with the Declaration of Helsinki and consent form will be obtained from the patients participating in the study, indicating that they are willing to participate in the study. Before starting the study, the purpose of the study will be explained to the participants and all information about the study will be provided. The subjects who agree to participate in the study will be invited to Istanbul University Faculty of Medicine, Department of Chest Diseases on certain days. Demographic information of the subjects will be recorded. Body composition, presence of comorbidities, exercise capacity, peripheral muscle strength, sleep quality and quality of life will then be assessed. The primary aim of the study was to investigate whether Obesity Hypoventilation Syndrome has an additional effect on exercise capacity, peripheral muscle strength and quality of life compared to obesity.

ELIGIBILITY:
Inclusion Criteria:

* 30 < body mass index < 45 kg/m2
* Patients who have been diagnosed with Obesity Hypoventilation Syndrome
* Obese subjects with low risk of obstructive sleep apnea (STOP-BANG score < 3)

Exclusion Criteria:

* Patients with uncontrollable respiratory and comorbid diseases
* Patient who have been an orthopedic, neurological, cardiac, or metabolic condition that may prevent participation and continuation of the exercise program throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Obesity Hypoventilation Syndrome who are followed up in Istanbul University, Istanbul Faculty of Medicine, Department of Chest Diseases and obese individuals who are followed up in Istanbul University, Istanbul Faculty of Medicine, Department of Internal Diseases and who are in the low risk group according to stop bang evaluation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test-Distance | 1 day
  The distance covered in meters in a straight corridor of 30 meters will be recorded as fast as possible but without running for 6 minutes.
Six Minute Walk Test-Oxygen Saturation | 1 day
  The 6-minute walk test is performed by walking as fast as possible for 6 minutes in a 30-meter corridor. Oxygen saturation measured by pulse oximetry before and after the test is recorded as a percentage.
Six Minute Walk Test-Heart Rate | 1 day
  The 6-minute walk test is performed by walking as fast as possible for 6 minutes in a 30-meter corridor. The heart rate measured by pulse oximetry is recorded before and after the test.
Six Minute Walk Test-Blood Pressure | 1 day
  The 6-minute walk test is performed by walking as fast as possible for 6 minutes in a 30-meter corridor. Before and after the test, blood pressure is measured with a sphygmomanometer and recorded in mmHg.
Six Minute Walk Test-Dyspnea | 1 day
  The 6-minute walk test is performed by walking as fast as possible for 6 minutes in a 30-meter corridor. Before and after the test, a score of 0-10 is recorded according to the Borg scale.
Six Minute Walk Test-Leg Fatigue | 1 day
  6 dakika yürüme testi, kişinin 30 metrelik bir koridorda 6 dakika boyunca mümkün olabilecek en hızlı şekilde yürümesi ile gerçekleştirilmektedir. Test öncesi ve sonrasında Borg skalasına göre 0-10 arasında puanlandırılarak kaydedilir.
Nottingham Health Profile | 1 day
  The Nottingham Health Profile (NHP) is a general patient reported outcome measure which seeks to measure subjective health status. It is a questionnaire designed to measure a patient's view of their own health status, in a number of areas. The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. The second part of the NHP is optional and can be omitted without ruining the test results.
Muscle Strength - Dynamometer | 1 day
  A digital dynamometer will be used to evaluate muscle strength. Muscle strength will be evaluated in the following muscles, each measurement will be made three times and the average will be taken.

SECONDARY OUTCOMES:
Body Fat Percentage | 1 day
  The body fat percentage of a patient is the total mass of fat divided by total body mass, multiplied by 100; body fat includes essential body fat and storage body fat. The body fat percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in percent.
Body Fluid Percentage | 1 day
  Body fluids, bodily fluids, or biofluids are liquids within the human body. The body fluid percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in percent.
Muscle Mass | 1 day
  Muscle mass refers to the amount of soft muscle tissue in the body. The muscle mass of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in kg.
Body Mass Index | 1 day
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Anthropometric Measurements-Neck | 1 day
  With the help of a tape measure, neck circumference will be measured in cm.
Anthropometric Measurements-Waist | 1 day
  With the help of a tape measure, waist circumference will be measured in cm.
Anthropometric Measurements-Abdomen | 1 day
  With the help of a tape measure, abdomen circumference will be measured in cm.
Anthropometric Measurements-Hip | 1 day
  With the help of a tape measure, hip circumference will be measured in cm.
The Waist-Hip ratio | 1 day
  With the help of a tape measure, waist and hip circumference will be measured in cm. Depending on the circumference measurements, waist and hip circumference is calculated as waist to hip ratio.
Modified Charlson Comorbidity Index | 1 day
  The Charlson Comorbidity Index (CCI) was initially developed to predict the survival time of individuals diagnosed with cancer by assigning weights to specific diseases. Today, it is used as a guide for individuals with multiple comorbidities. In this index, diseases are scored based on their morbidity and mortality. The total score is calculated by summing the equivalent scores of diseases. Comorbidity classification is categorized as low (score ≤ 3), moderate (score 4 and 5), high (score 6 and 7), and very high comorbidity (score ≥ 8).
Pittsburgh Sleep Quality Index | 1 day
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Goksen KURAN ASLAN, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa; Ece ACIKBAS, PT,MSc, Study Chair — Istanbul University - Cerrahpasa; Ozge ERTAN HARPUTLU, PT,MSc, Study Chair — Istanbul University - Cerrahpasa; Esen KIYAN, Prof, Study Chair — Istanbul University; Bedia Fulya CALIKOGLU, Lect. PhD, Study Chair — Istanbul University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No